CLINICAL TRIAL: NCT03887572
Title: Getting Older Patients Walking: Adaption of MOVIN (Mobilizing Older Adult Patients Via a Systems-based INtervention) for Implementation in a Non-Academic Hospital
Brief Title: Adaption of Mobilizing Older Adult Patients Via a Systems-based Intervention for a Non-Academic Hospital
Acronym: MOVIN
Status: Completed | Type: Observational
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: Wake Forest University Health Sciences (Other); National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Other Study IDs: 2018-1025; A545000 (Other: UW Madison); NUR/FACULTY AFFAIRS/ADMIN (Other: UW Madison); 1UL1TR002373-01 (NIH)
Record Dates: First submitted 2019-03-14; First posted 2019-03-25 (Actual); Last update posted 2024-04-19 (Actual); Status verified 2024-04

CONDITIONS: Early Mobility; Older Adults; Hospital Acquired Condition
MeSH Terms: conditions — Iatrogenic Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Pre-intervention/control: 20 older adult patients (age 65 or older) will be recruited over 3 months prior to implementation of the unit-based MOVIN intervention.
- Post-intervention: 20 older adult patients (age 65 or older) will be recruited over 3 months after MOVIN has been implemented on the unit for a period of 12-14 weeks.
  Interventions: Other: MOVIN

INTERVENTIONS:
Other: MOVIN — MOVIN is a multi-component unit-based intervention comprised of five components that are implemented simultaneously in a hospital unit. The five components are: 1) psychomotor skills training, 2) unit ambulation culture, 3) communication, 4) resources, 5) ambulation environment.
  Groups: Post-intervention

SUMMARY:
This observational study is designed to adapt, create actionable implementation, and to access market demand of the Mobilizing Older adults Via a systems-based Intervention (MOVIN) toolkit. MOVIN is a program to increase ambulation while hospitalized at non-academic facilities. MOVIN is a unit-based intervention. Therefore all patients on this unit are exposed to the intervention once it is implemented regardless of whether or not they participate in the trial. The study will enroll 40 total hospitalized participants 65 years and older for the duration of their stay.

DETAILED DESCRIPTION:
Up to 65% of hospitalized older adults will lose the ability to ambulate independently during their hospital stay. Loss of independent ambulation has been identified as a hospital-acquired disability and is a critical patient safety concern, resulting in permanent loss of function for 50% of older adults one-year post discharge. Functional loss is associated with multiple negative outcomes including a 33% increase in new nursing home placement, increase in length of hospital stay, need for home health services, falls, caregiver burden, decreased quality of life, and increased mortality. Given the rapid increase in the elderly population, loss of independent ambulation primarily due to the process of care in hospital settings may significantly increase future healthcare costs and further exacerbate concerns related to patient care quality.

Lack of walking during hospitalization has been directly linked to loss of independent ambulation in older adults. Nurses are responsible for promoting and maintaining patient independent mobility. However, our research has identified multiple personal and organizational barriers that prevent nurses from walking patients. We have developed and pilot tested a novel systems based multi-component intervention to improve ambulation of older adult patients, Mobilizing Older adult patients Via a systems-based INtervention (MOVIN). MOVIN is comprised of five components: 1) psychomotor skills training; 2) communication tools; 3) ambulation pathways; 4) ambulation resources; and 5) unit ambulation culture. Our pilot study of MOVIN demonstrated a statistically significant increase in frequency and weekly distance of patient ambulation as well as changes in nursing practice and unit culture. Notably, these changes have been sustained for greater than two years after completion of the study.

Our goal is to translate our positive research results into an actionable implementation package that can be used to disseminate MOVIN to hospitals nationwide and improve the quality of care and functional outcomes for older adult patients. In pursuit of this goal, our specific aims are to:

1. Adapt MOVIN and develop and refine a MOVIN toolkit for implementation in a non-academic hospital.
2. Implement MOVIN in an inpatient adult general medical unit in a non-academic hospital with an on-site clinical team leading the intervention and evaluate using the RE-AIM framework to collect preliminary data for a future dissemination study.
3. Assess market demand for the intervention and develop a customer value statement in collaboration with the ICTR Dissemination and Implementation Program.

ELIGIBILITY:
Inclusion Criteria:

* age 65 years or older
* able to walk with or without assistance
* absence of a medical order for bedrest or activity restriction
* have an ambulation order
* able to speak and understand English.

Exclusion Criteria:

* activated Power of Attorney
* a score of 11+ on Orientation Memory Cognition Test (OMCT)
* a score <2 on a Mini Cog
* lower extremity amputation
* terminal diagnosis (Comfort Care)
* on hospice
* bed rest order
* wheelchair bound

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patients admitted to the study intervention unit will be recruited to evaluate the implementation of MOVIN based on Reach, Effectiveness, Adoption, Implementation and Maintenance (RE-AIM framework). Patients (N=40) will be recruited during pre (n=20) and post (n=20)-intervention periods to provide an evaluation of effectiveness. Inclusion criteria for patients will consist of age 65 years or older, able to walk with or without assistance, have an ambulation order, and able to speak and understand English.
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2019-03-04 (Actual); Primary Completion 2020-02-04 (Actual); Study Completion 2020-02-04 (Actual)

PRIMARY OUTCOMES:
Change in gait speed | Hospital admission, hospital discharge, 3 months post-discharge; Up to 4 months total
  A 4 meter walk test will be conducted on admission to the study, discharge from the hospital and at 3 months post discharge in the subjects home or the hospital or clinic. A trained member of the research team will conduct the gait speed test. Interrater reliability for the 4 meter walk test will be conducted between all members of the research team prior to collecting gait speed data on study participants. Gait Speed is a physical performance measure identified as a sensitive clinical indicator of health, mortality, healthcare utilization, and independence in ambulation, and is feasible to test in hospitalized older adults. Change scores will be calculated as the difference between gait speeds measured at each of these time points.
Change in Self-report on Katz Activity of Daily Living (ADL) Index | Hospital admission, hospital discharge, 1 month post-discharge, 3 months post-discharge; Up to 4 months total
  A trained member of the research team will collect patients self-report of ADLs on admission to the study, discharge from the hospital, by phone at 1 month post intervention, and in person at the 3 month post intervention visit. The Katz ADL Index is a self-report scale that measures five ADL on three levels (independent, requiring assistance of another and unable to do). The scale demonstrates excellent reliability and predictive validity, and is sensitive to change in hospital settings. Change scores will be calculated as the difference between gait speeds measured at each of these time points.
Change in Life Space Assessment | Hospital admission, hospital discharge, 1 month post-discharge, 3 months post-discharge; Up to 4 months total
  A trained member of the research team will collect patients self-report on Life Space at admission to the study, discharge from the hospital, by phone at 1 month post intervention, and in person at the 3 month post intervention visit. The UAB Life Space Assessment: is a self-report scale of ambulation that measures spaces patients' move in, the frequency of moving into those spaces, and dependency in moving into those spaces. This scale has demonstrated reliability and predictive validity and sensitivity to change after hospital stay. Change scores will be calculated as the difference between gait speeds measured at each of these time points.

SECONDARY OUTCOMES:
Patient Experience with Ambulation | 1 month post-discharge; Up to 2 months total
  Brief interviews will be conducted to further examine and understand the patient experience with ambulation on the inpatient unit.
Age | Within 3 months post-discharge; Up to 4 months total
  Age in years will be collected via patient medical record review by a nurse researcher from the study team.
Gender | Within 3 months post-discharge; Up to 4 months total
  Gender will be collected via patient medical record review by a nurse researcher from the study team
Race | Within 3 months post-discharge; Up to 4 months total
  Race will be collected via patient medical record review by a nurse researcher from the study team.
Ethnicity | Within 3 months post-discharge; Up to 4 months total
  Ethnicity will be collected via patient medical record review by a nurse researcher from the study team.
Social support | Post-discharge; Up to 1 month
  Social support (defined as: living alone, living with another, presence of a caregiver, use of home care services) will be collected via patient medical record review by a nurse researcher from the study team.
Location admitted from | Within 3 months post-discharge; Up to 4 months total
  Location admitted from (defined as: home, assisted living, nursing home, other hospital, other inpatient unit) will be collected via patient medical record review by a nurse researcher from the study team.
Reason for admission | Within 3 months post-discharge; Up to 4 months total
  Reason for admission will be collected via patient medical record review by a nurse researcher from the study team.
Use of an ambulation assistive device | Within 3 months post-discharge; Up to 4 months total
  Use of an ambulation assistive device (including, walker, cane, wheelchair) will be collected via patient medical record review by a nurse researcher from the study team.
Presence of external lines | Within 3 months post-discharge; Up to 4 months total
  Presence of external lines (Foley catheter, intravenous lines, supplemental oxygen, drainage tubes) will be collected via patient medical record review by a nurse researcher from the study team.
Body Mass Index | Within 3 months post-discharge; Up to 4 months total
  Body Mass Index will be collected via patient medical record review by a nurse researcher from the study team.
Fall risk | Within 3 months post-discharge; Up to 4 months total
  Documentation of fall risk status will be collected via patient medical record review by a nurse researcher from the study team.
Fall reported | Within 3 months post-discharge; Up to 4 months total
  Whether or not a fall was reported during the hospital stay will be collected via patient medical record review by a nurse researcher from the study team.
Length of stay | Within 3 months post-discharge; Up to 4 months total
  Length of hospital stay will be collected via patient medical record review by a nurse researcher from the study team.
Discharge destination | Within 3 months post-discharge; Up to 4 months total
  Discharge destination (home, skilled nursing facility) will be collected via patient medical record review by a nurse researcher from the study team.
Charlson Comorbidity Index | Within 3 months post-discharge; Up to 4 months total
  This index will be calculated via chart review by a nurse researcher member of the study team.

CONTACTS AND LOCATIONS:
Overall Officials: Linsey M Steege, PhD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- Aurora St. Luke's Medical Center, Milwaukee, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No